CLINICAL TRIAL: NCT03934541
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of an HIV-1 gp41 MPER-656 Liposome Vaccine in Healthy, HIV-uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of an HIV-1 gp41 MPER-656 Liposome Vaccine in Healthy, HIV-uninfected Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 133; 12047 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Treatment 1): MPER-656 Liposome Vaccine (Experimental): Participants will receive 500 mcg of MPER-656 liposomes, admixed with Aluminum Hydroxide Suspension, to be administered as two 0.5 mL doses at Months 0, 2, and 6.
  Interventions: Biological: MPER-656 Liposome Vaccine
- Group 1 (Control 1): Placebo for MPER-656 Liposome Vaccine (Placebo Comparator): Participants will receive placebo to be administered as two 0.5 mL doses at Months 0, 2, and 6.
  Interventions: Biological: Placebo for MPER-656 Liposome Vaccine
- Group 2 (Treatment 2): MPER-656 Liposome Vaccine (Experimental): Participants will receive 2000 mcg of MPER-656 liposomes, admixed with Aluminum Hydroxide Suspension, to be administered as two 0.5 mL doses at Months 0, 2, and 6.
  Interventions: Biological: MPER-656 Liposome Vaccine
- Group 2 (Control 2): Placebo for MPER-656 Liposome Vaccine (Placebo Comparator): Participants will receive placebo to be administered as two 0.5 mL doses at Months 0, 2, and 6.
  Interventions: Biological: Placebo for MPER-656 Liposome Vaccine

INTERVENTIONS:
Biological: MPER-656 Liposome Vaccine — Administered by intramuscular injection
  Arms: Group 1 (Treatment 1): MPER-656 Liposome Vaccine; Group 2 (Treatment 2): MPER-656 Liposome Vaccine
Biological: Placebo for MPER-656 Liposome Vaccine — Administered by intramuscular injection
  Arms: Group 1 (Control 1): Placebo for MPER-656 Liposome Vaccine; Group 2 (Control 2): Placebo for MPER-656 Liposome Vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of an HIV-1 gp41 MPER-656 liposome vaccine in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of an HIV-1 gp41 MPER-656 liposome vaccine in healthy, HIV-uninfected adults.

Participants will be randomly assigned to four groups. Participants in Group 1 (Treatment 1) will receive 500 mcg of MPER-656 liposome vaccine at Months 0, 2, and 6. Participants in Group 1 (Control 1) will receive placebo at Months 0, 2, and 6. Participants in Group 2 (Treatment 2) will receive 2000 mcg of MPER-656 liposome vaccine at Months 0, 2, and 6. Participants in Group 2 (Control 2) will receive placebo at Months 0, 2, and 6. Study staff will review safety data from Group 1 before deciding whether to enroll Group 2.

Participants will attend several study visits through Month 12. Visits may include physical examinations, blood and urine collection, HIV testing, risk reduction counseling, and questionnaires. Study staff will contact participants at Month 18 for follow-up health monitoring.

As of May 2020, vaccinations were discontinued for all participants.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent while in this study
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see study protocol for more information)

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth)
* White blood cell count equal to 2,500 to 12,000 cells/mm^3 with normal differential, or differential approved by Investigator of Record (IoR) as not clinically significant
* Total lymphocyte count greater than or equal to 650 cells/mm^3 with normal differential, or differential approved by IoR as not clinically significant
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000 cells/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to 1.1 times the institutional upper limit of normal

Clotting and autoantibodies

* Anticardiolipin IgG antibodies below the upper limit of normal
* Negative antinuclear antibodies

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative FDA-approved enzyme immunoassay (EIA)
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative or trace urine protein, and
  * Negative, trace, or 1+ blood urine hemoglobin (if +1 hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range)

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test at screening (ie, prior to randomization) and prior to study product administration on the day of study product administration. Persons who are NOT of reproductive potential due to having undergone hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth:

  * Must agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit
  * Effective contraception is defined as using the following methods:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception,
    * Tubal ligation, or
    * Any other contraceptive method approved by the HVTN 133 Protocol Safety Review Team (PSRT),
    * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, or bilateral oophorectomy,
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 133 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 133 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 133 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 1 year in a prior vaccine trial. Exceptions may be made by the HVTN 133 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 133 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 1 year ago, eligibility for enrollment will be determined by the HVTN 133 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than or equal to 60 mg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment)
* Serious adverse reactions to vaccines or to vaccine components including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination (for mAb see criterion above)
* Autoimmune disease, current or history, (Not exclusionary: mild, wellcontrolled psoriasis)
* Adverse event of special interest (AESIs): Volunteers who currently have, or have a history of any condition that could be considered an AESI for the products administered in this protocol (representative examples are listed in the study protocol)
* Immunodeficiency

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Any contraindication that would preclude injections into both left and right deltoids
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria: Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has had either of the following:

    * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2. (Not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months (Not exclusionary: well-controlled non-autoimmune thyroid disease)
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently less than 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of generalized urticaria, angioedema, or anaphylaxis. (Not exclusionary: angioedema or anaphylaxis to a known trigger with at least 5 years since last reaction to demonstrate satisfactory avoidance of trigger.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, Study Chair — Brigham and Women's Hospital; Nathan Erdmann, Study Chair — University of Alabama at Birmingham
Locations (6):
- United States (6):
  - Alabama CRS, Birmingham, Alabama
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Derived] Erdmann N, Williams WB, Walsh SR, Cain DW, Clark M, Tuck R, Holmes S, Clardy B, Foulger A, Parks R, Barr M, Eaton A, Saunders KO, Grunenberg N, Edlefsen P, Goepfert PA, Cohen KW, Maenza J, Mayer K, Van Tieu H, Sobieszczyk ME, Swann E, Lu H, De Rosa SC, Sagawa ZK, Lin BC, Carrol RE, McKee K, Doria-Rose NA, Louder MK, Moody MA, Fox CB, Ferrari G, Edwards RJ, Acharya P, Alam SM, Tomaras GD, Montefiori DC, Gilbert PB, McElrath MJ, Corey L, Haynes BF, Baden LR; NIAID HVTN 133 Study Group. An HIV-1 gp41 peptide-liposome vaccine elicits neutralizing epitope-targeted antibody responses in healthy individuals. medRxiv [Preprint]. 2025 Aug 22:2024.03.15.24304305. doi: 10.1101/2024.03.15.24304305. PMID 38562833

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1: 500 mcg MPER-656 mo(0,2,6,12): MPER-656 liposomes, 500 mcg, admixed with Aluminum Hydroxide Suspension, to be administered as two 0.5 mL doses intramuscularly (IM) at months 0, 2, 6, and 12.
- Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12): MPER-656 liposomes, 2000 mcg, admixed with Aluminum Hydroxide Suspension, to be administered as two 0.5 mL doses IM at months 0, 2, 6, and 12.
- Control 1: Placebo for MPER-656 mo(0,2,6,12); Control 2: Placebo for MPER-656 mo(0,2,6,12): Placebo for MPER-656 liposomes (Sodium Chloride for Injection USP, 0.9%) to be administered as two 0.5 mL doses IM at months 0, 2, 6, and 12.
Period: Overall Study
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Started | 5 | 15 | 1 | 3
Completed | 5 | 14 | 1 | 3
Not Completed | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12) | Total
Number analyzed (Participants) | 5 | 15 | 1 | 3 | 24
Age, Continuous [Median (Full Range); unit: years] | 24 [21 to 33] | 29 [18 to 37] | 30 [30 to 30] | 23 [22 to 40] | 27 [18 to 40]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 0 | 1 | 0 | 0 | 1
  21 - 30 years | 3 | 7 | 1 | 2 | 13
  31 - 40 years | 2 | 7 | 0 | 1 | 10
  41 - 50 years | 0 | 0 | 0 | 0 | 0
  Above 50 years | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 12 | 0 | 2 | 16
  Male | 3 | 3 | 1 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 15 | 1 | 2 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 4 | 11 | 1 | 2 | 18
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 15 | 1 | 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through 7 days after each vaccine dose at Months (0,2,6,12)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Participants
  None | 1 | 0 | 1 | 3
  Mild | 2 | 11 | 0 | 0
  Moderate | 2 | 4 | 0 | 0
  Severe | 0 | 0 | 0 | 0
  Potentially life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 7 days after each vaccine dose at Months (0,2,6,12)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Participants
  Erythema/redness: None | 3 | 14 | 1 | 3
  Erythema/redness: Not Gradable | 1 | 1 | 0 | 0
  Erythema/redness: Gr 1: 2.5 to less than 5 cm dim. | 0 | 0 | 0 | 0
  Erythema/redness: Gr 2: 5 to less than 10 cm dim. | 0 | 0 | 0 | 0
  Erythema/redness: Gr 3: >=10 cm dim. | 1 | 0 | 0 | 0
  Erythema/redness: Gr 3: Complications AE | 0 | 0 | 0 | 0
  Erythema/redness: Gr 4: Complications AE | 0 | 0 | 0 | 0
  Induration/swelling: None | 3 | 12 | 1 | 3
  Induration/swelling: Not Gradable | 1 | 1 | 0 | 0
  Induration/swelling: Gr 1: 2.5 to less than 5 cm dim. | 0 | 2 | 0 | 0
  Induration/swelling: Gr 2: 5 to less than 10 cm dim. | 0 | 0 | 0 | 0
  Induration/swelling: Gr 3: >=10 cm dim. | 1 | 0 | 0 | 0
  Induration/swelling: Gr 3: Complications AE | 0 | 0 | 0 | 0
  Induration/swelling: Gr 4: Complications AE | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 2 | 12 | 1 | 3
  Erythema and/or Induration: Not Gradable | 2 | 1 | 0 | 0
  Erythema and/or Induration: Gr 1: 2.5 to less than 5 cm dim. | 0 | 2 | 0 | 0
  Erythema and/or Induration: Gr 2: 5 to less than 10 cm dim. | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 3: >=10 cm dim. | 1 | 0 | 0 | 0
  Erythema and/or Induration: Gr 3: Complications AE | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 4: Complications AE | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities excluding body temperature for a participant.
Time Frame: Measured through 7 days after each vaccine dose at Months (0,2,6,12)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Participants
  Arthralgia: None | 3 | 13 | 1 | 3
  Arthralgia: Mild | 2 | 2 | 0 | 0
  Arthralgia: Moderate | 0 | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0
  Arthralgia: Potentially life-threatening | 0 | 0 | 0 | 0
  Chills: None | 4 | 14 | 1 | 2
  Chills: Mild | 1 | 1 | 0 | 1
  Chills: Moderate | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0
  Chills: Potentially life-threatening | 0 | 0 | 0 | 0
  Headache: None | 3 | 9 | 1 | 1
  Headache: Mild | 2 | 5 | 0 | 2
  Headache: Moderate | 0 | 1 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0
  Headache: Potentially life-threatening | 0 | 0 | 0 | 0
  Malaise and/or fatigue: None | 1 | 8 | 1 | 2
  Malaise and/or fatigue: Mild | 4 | 5 | 0 | 1
  Malaise and/or fatigue: Moderate | 0 | 2 | 0 | 0
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 10 | 1 | 3
  Myalgia: Mild | 2 | 4 | 0 | 0
  Myalgia: Moderate | 0 | 1 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Myalgia: Potentially life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 4 | 10 | 1 | 2
  Nausea: Mild | 1 | 5 | 0 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Potentially life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 1 | 3 | 1 | 1
  Max. Systemic Symptoms: Mild | 4 | 9 | 0 | 2
  Max. Systemic Symptoms: Moderate | 0 | 3 | 0 | 0
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially life-threatening | 0 | 0 | 0 | 0
  Temperature (C): None | 5 | 15 | 1 | 3
  Temperature (C): Mild | 0 | 0 | 0 | 0
  Temperature (C): Moderate | 0 | 0 | 0 | 0
  Temperature (C): Severe | 0 | 0 | 0 | 0
  Temperature (C): Potentially life-threatening | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT) in U/L
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during screening, Days 14, 70, 182
Population: Overall Number of Participants Analyzed represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
U/L
  Alanine Aminotransferase (U/L)-Baseline | 14 [13 to 20] | 15 [11 to 20] | 17 [17 to 17] | 14 [11 to 17]
  Alanine Aminotransferase (U/L)-Day 14 | 21 [10 to 23] | 11 [10 to 19] | 15 [15 to 15] | 12 [8 to 14]
  Alanine Aminotransferase (U/L)-Day 70 | 14 [11 to 27] | 14 [11 to 16] | 15 [15 to 15] | 9 [9 to 13]
  Alanine Aminotransferase (U/L)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Alanine Aminotransferase (U/L)-Day 182 | 19 [13.5 to 40.5] | 16 [14 to 18] | 16 [16 to 16] | 13 [13 to 13]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine in mg/dL
Description: as for outcome 4
Time Frame: Measured during screening, Days 14, 70, 182
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
mg/dL
  Creatinine (mg/dL)-Baseline | 0.97 [0.78 to 1] | 0.73 [0.7 to 0.85] | 0.68 [0.68 to 0.68] | 0.7 [0.69 to 0.81]
  Creatinine (mg/dL)-Day 14 | 1 [0.96 to 1.07] | 0.7 [0.67 to 0.8] | 0.74 [0.74 to 0.74] | 0.82 [0.63 to 0.96]
  Creatinine (mg/dL)-Day 70 | 0.92 [0.9 to 1.01] | 0.72 [0.65 to 0.8] | 0.76 [0.76 to 0.76] | 0.83 [0.74 to 0.93]
  Creatinine (mg/dL)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Creatinine (mg/dL)-Day 182 | 0.88 [0.82 to 0.96] | 0.78 [0.75 to 0.81] | 0.82 [0.82 to 0.82] | 0.71 [0.71 to 0.71]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin in g/dL
Description: as for outcome 4
Time Frame: Measured during screening, Days 14, 70, 182
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
g/dL
  Hemoglobin (g/dL)-Baseline | 14 [13 to 16] | 14 [13 to 14] | 14 [14 to 14] | 14 [12 to 15]
  Hemoglobin (g/dL)-Day 14 | 13 [13 to 15] | 13 [12 to 14] | 13 [13 to 13] | 13 [11 to 13]
  Hemoglobin (g/dL)-Day 70 | 13 [13 to 15] | 13 [12 to 14] | 15 [15 to 15] | 12 [11 to 14]
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Hemoglobin (g/dL)-Day 182 | 14 [13 to 15] | 12 [12 to 13] | 14 [14 to 14] | 14 [14 to 14]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: Measured during screening, Days 14, 70, 182
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
1000 cells/cubic mm
  Lymphocytes (1000 cells/cubic mm)-Baseline | 2.44 [2.2 to 2.508] | 2.09 [1.84 to 2.227] | 2.39 [2.39 to 2.39] | 2.587 [2.335 to 2.7]
  Lymphocytes (1000 cells/cubic mm)-Day 14 | 2.25 [1.84 to 2.677] | 2.027 [1.77 to 2.563] | 1.87 [1.87 to 1.87] | 1.876 [1.626 to 3.14]
  Lymphocytes (1000 cells/cubic mm)-Day 70 | 2.27 [2.04 to 2.391] | 2.017 [1.81 to 2.5] | 1.88 [1.88 to 1.88] | 1.811 [1.793 to 2.48]
  Lymphocytes (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Lymphocytes (1000 cells/cubic mm)-Day 182 | 2.53 [2.405 to 3.085] | 2.335 [1.68 to 2.99] | 1.77 [1.77 to 1.77] | 2.67 [2.67 to 2.67]
  Neutrophils (1000 cells/cubic mm)-Baseline | 4.42 [3.05 to 4.68] | 3.79 [2.96 to 4.61] | 4.48 [4.48 to 4.48] | 5.216 [4.612 to 6.14]
  Neutrophils (1000 cells/cubic mm)-Day 14 | 3.99 [3 to 4.12] | 3.76 [2.9 to 4.76] | 1.99 [1.99 to 1.99] | 5.7 [4.963 to 8.238]
  Neutrophils (1000 cells/cubic mm)-Day 70 | 3.8 [2.94 to 4.12] | 3.47 [2.808 to 5.39] | 1.55 [1.55 to 1.55] | 5.412 [4.757 to 6.33]
  Neutrophils (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Neutrophils (1000 cells/cubic mm)-Day 182 | 4.135 [3.77 to 4.89] | 3.93 [2.97 to 4.89] | 1.91 [1.91 to 1.91] | 5.78 [5.78 to 5.78]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, WBC in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: Measured during screening, Days 14, 70, 182
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
1000 cells/cubic mm
  WBC (1000 cells/cubic mm)-Baseline | 7.61 [6.37 to 9] | 6.51 [5.9 to 7.44] | 7.6 [7.6 to 7.6] | 8.4 [7.7 to 9.47]
  WBC (1000 cells/cubic mm)-Day 14 | 7.28 [6.53 to 8.01] | 6.54 [5.2 to 7.56] | 4.53 [4.53 to 4.53] | 9.83 [7.1 to 11.3]
  WBC (1000 cells/cubic mm)-Day 70 | 6.93 [5.76 to 7.27] | 6.38 [5.26 to 8.77] | 4.04 [4.04 to 4.04] | 8.3 [7.1 to 9.61]
  WBC (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  WBC (1000 cells/cubic mm)-Day 182 | 7.91 [7.37 to 8.66] | 7.12 [5.41 to 8.83] | 4.32 [4.32 to 4.32] | 9.19 [9.19 to 9.19]
  Platelets (1000 cells/cubic mm)-Baseline | 229 [218.8 to 235] | 250 [220.2 to 323] | 242 [242 to 242] | 290 [267 to 294]
  Platelets (1000 cells/cubic mm)-Day 14 | 218 [211 to 264] | 277 [240 to 347.9] | 227 [227 to 227] | 306 [288 to 353]
  Platelets (1000 cells/cubic mm)-Day 70 | 237 [197.6 to 279] | 278 [235.6 to 326.1] | 260 [260 to 260] | 298 [282 to 325]
  Platelets (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Platelets (1000 cells/cubic mm)-Day 182 | 235.8 [212.8 to 256] | 285.5 [219 to 352] | 231 [231 to 231] | 317 [317 to 317]

9. Primary Outcome: The Number (Percentage) of Participants With Lab Grade > 1 for Alanine Aminotransferase (ALT), Creatinine, Hemoglobin, Lymphocyte Count, Neutrophil Count, Platelets, White Blood Cells (WBC) Was Summarized by Arm
Description: The number (percentage) of participants with lab grade > 1 for alanine aminotransferase (ALT), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by arm.
Time Frame: Measured during screening, Days 14, 70, 182
Population: Overall Number of Participants Analyzed represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Participants
  Alanine Aminotransferase (U/L)-Baseline | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 14 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 70 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Alanine Aminotransferase (U/L)-Day 182 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Baseline | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 14 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 70 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Hemoglobin (g/dL)-Day 182 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Baseline | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 14 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 70 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Creatinine (mg/dL)-Day 182 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 14 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 70 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  WBC (1000 cells/cubic mm)-Day 182 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 14 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 70 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Platelets (1000 cells/cubic mm)-Day 182 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 14 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 70 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Lymphocytes (1000 cells/cubic mm)-Day 182 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 14 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 70 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 182: number analyzed (Participants) | 4 | 2 | 1 | 1
  Neutrophils (1000 cells/cubic mm)-Day 182 | 0 | 0 | 0 | 0

10. Primary Outcome: Occurrence and Level of MPER-peptide-specific IgG Binding Ab Responses as Assessed by Binding Ab Multiplex Assay With MPER-656 Liposome Vaccine - Response Rates
Description: Serum HIV-1-specific IgG responses against antigens listed below were on a Bio-Plex instrument (Bio-Rad) using a standardized custom HIV-1 Luminex assay, run at 1:50 dilution. The readout was background-subtracted mean fluorescence intensity (MFI), where background referred to a plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen minus reference antigen MFI. Net MFI below 1 is set to 1, and Net MFI above 22,000 is set to 22,000. Samples from post-baseline visits have positive responses if they meet three criteria: (1) net MFI >= antigen-specific threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI > 3 times baseline net MFI, and (3) experimental antigen MFI > 3 times baseline MFI. Data are excluded if the blood draw date was outside the allowable window, a participant was HIV-infected, or the reference antigen exceeds 6500 MFI.
Time Frame: Measured at Month 2.5(V5) and Month 6.5(V7)
Population: Avaiable Data at V5 and V7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Participants
  IgG - Clade C MPER - Month 2.5(V5) | 0 | 0 | 0 | 0
  IgG - Clade C MPER - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - Clade C MPER - Month 6.5(V7) | 0 | 0 | 0 | 0
  IgG - NA/MPER656-GTH1-biotin - Month 2.5(V5) | 5 | 14 | 0 | 0
  IgG - NA/MPER656-GTH1-biotin - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - NA/MPER656-GTH1-biotin - Month 6.5(V7) | 3 | 1 | 0 | 0
  IgG - SP62 - Month 2.5(V5) | 5 | 15 | 0 | 0
  IgG - SP62 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - SP62 - Month 6.5(V7) | 3 | 1 | 0 | 0
  IgG - gp41 - Month 2.5(V5): number analyzed (Participants) | 5 | 14 | 1 | 3
  IgG - gp41 - Month 2.5(V5) | 2 | 12 | 0 | 0
  IgG - gp41 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - gp41 - Month 6.5(V7) | 2 | 1 | 0 | 0

11. Primary Outcome: Occurrence and Level of MPER-peptide-specific IgG Binding Ab Responses as Assessed by Binding Ab Multiplex Assay With MPER-656 Liposome Vaccine - Magnitudes
Description: as for outcome 10
Time Frame: Measured at Month 2.5(V5) and Month 6.5(V7)
Population: Avaiable Data at V5 and V7
Measure: Median (Inter-Quartile Range); unit: Relative luminescence units (RLU)
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Relative luminescence units (RLU)
  IgG - Clade C MPER - Month 2.5(V5) | 6.25 [3.5 to 16] | 4.75 [1.75 to 10.38] | 7.75 [7.75 to 7.75] | 1 [1 to 1]
  IgG - Clade C MPER - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - Clade C MPER - Month 6.5(V7) | 5.38 [3.81 to 7.81] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  IgG - NA/MPER656-GTH1-biotin - Month 2.5(V5) | 8714.25 [4366.75 to 17715] | 21821.75 [10803.62 to 22000] | 11 [11 to 11] | 20.5 [14.62 to 216.62]
  IgG - NA/MPER656-GTH1-biotin - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - NA/MPER656-GTH1-biotin - Month 6.5(V7) | 17438.62 [9718.19 to 22000] | 22000 [22000 to 22000] | 11.75 [11.75 to 11.75] | 660.5 [660.5 to 660.5]
  IgG - SP62 - Month 2.5(V5) | 1057.5 [883.75 to 3674] | 2593 [1052.75 to 5125.5] | 12 [12 to 12] | 1.75 [1.38 to 5.88]
  IgG - SP62 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - SP62 - Month 6.5(V7) | 6435.5 [937.69 to 13783.44] | 3753.5 [3753.5 to 3753.5] | 8.25 [8.25 to 8.25] | 1 [1 to 1]
  IgG - gp41 - Month 2.5(V5) | 765.5 [716.25 to 4287.75] | 1879.75 [993.12 to 5622.38] | 678 [678 to 678] | 384.25 [245.5 to 421.75]
  IgG - gp41 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  IgG - gp41 - Month 6.5(V7) | 5806.5 [580.81 to 13653.81] | 2974.25 [2974.25 to 2974.25] | 565 [565 to 565] | 139 [139 to 139]

12. Secondary Outcome: Occurrence and Level of TZM-bl Cells Responses Against HIV-1 Viral Isolates - Response Rates
Description: Neutralizing antibodies against HIV-1 were measured as a function of reductions in Tat-regulated luciferase (Luc) reporter gene expression in TZM-bl and TZM-bl/Fcg RI cells . Assays in both cell lines measured neutralization titers as a function of a reduction in Tat-induced luciferase reporter gene expression after a single round of infection with Env-pseudotyped viruses. Test samples were assayed against a panel of HIV-1 strains that exhibit heightened susceptible to neutralization by MPER bnAbs in TZM-bl/Fcg RI cells.
Time Frame: Measured at Month 2.5(V5) and Month 6.5(V7)
Population: Avaiable Data at V5 and V7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Participants
  ID-50 - HXB2 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-50 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - HXB2 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-50 - SC422661.8 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-50 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - SC422661.8 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-50 - W61D(TCLA).71 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-50 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - W61D(TCLA).71 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-80 - HXB2 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-80 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - HXB2 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-80 - SC422661.8 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-80 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - SC422661.8 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-80 - W61D(TCLA).71 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-80 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - W61D(TCLA).71 - Month 6.5(V7) | 0 | 0 | 0 | 0

13. Secondary Outcome: Occurrence and Level of TZM-bl Cells Responses Against HIV-1 Viral Isolates - Magnitudes
Description: as for outcome 12
Time Frame: Measured at Month 2.5(V5) and Month 6.5(V7)
Population: Avaiable Data at V5 and V7
Measure: Median (Inter-Quartile Range); unit: Relative luminescence units (RLU)
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Relative luminescence units (RLU)
  ID-50 - HXB2 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - HXB2 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - SC422661.8 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - SC422661.8 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - W61D(TCLA).71 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - W61D(TCLA).71 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - HXB2 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - HXB2 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - SC422661.8 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - SC422661.8 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - W61D(TCLA).71 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - W61D(TCLA).71 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.

14. Secondary Outcome: Occurrence and Level of TZMbl/FcgRI Cells Responses Against HIV-1 Viral Isolates - Response
Description: as for outcome 12
Time Frame: Measured at Month 2.5(V5) and Month 6.5(V7)
Population: Avaiable Data at V5 and V7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Participants
  ID-50 - HXB2 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-50 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - HXB2 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-50 - SC422661.8 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-50 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - SC422661.8 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-50 - W61D(TCLA).71 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-50 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - W61D(TCLA).71 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-80 - HXB2 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-80 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - HXB2 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-80 - SC422661.8 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-80 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - SC422661.8 - Month 6.5(V7) | 0 | 0 | 0 | 0
  ID-80 - W61D(TCLA).71 - Month 2.5(V5) | 0 | 0 | 0 | 0
  ID-80 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - W61D(TCLA).71 - Month 6.5(V7) | 0 | 0 | 0 | 0

15. Secondary Outcome: Occurrence and Level of TZMbl/FcgRI Cells Responses Against HIV-1 Viral Isolates - Magnitudes
Description: as for outcome 12
Time Frame: Measured at Month 2.5(V5) and Month 6.5(V7)
Population: Avaiable Data at V5 and V7
Measure: Median (Inter-Quartile Range); unit: Relative luminescence units (RLU)
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
Number analyzed (Participants) | 5 | 15 | 1 | 3
Relative luminescence units (RLU)
  ID-50 - HXB2 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - HXB2 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - SC422661.8 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - SC422661.8 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - W61D(TCLA).71 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-50 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-50 - W61D(TCLA).71 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - HXB2 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - HXB2 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - HXB2 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - SC422661.8 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - SC422661.8 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - SC422661.8 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - W61D(TCLA).71 - Month 2.5(V5) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.
  ID-80 - W61D(TCLA).71 - Month 6.5(V7): number analyzed (Participants) | 4 | 1 | 1 | 1
  ID-80 - W61D(TCLA).71 - Month 6.5(V7) | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection. | NA [NA to NA] — Titers were below the level of detection.

ADVERSE EVENTS:
Time Frame: Serious adverse events of more than 30 days were collected through month 12. All other AEs were collected through 30 days after each vaccination (vaccinations were given at Months 0, 2, 6,12).
Arm/Group | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) | Control 1: Placebo for MPER-656 mo(0,2,6,12) | Control 2: Placebo for MPER-656 mo(0,2,6,12)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/15 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 4/5 | 10/15 | 0/1 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) (N=5) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) (N=15) | Control 1: Placebo for MPER-656 mo(0,2,6,12) (N=1) | Control 2: Placebo for MPER-656 mo(0,2,6,12) (N=3)
Any Event in SOC (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1: 500 mcg MPER-656 mo(0,2,6,12) (N=5) | Treatment 2: 2000 mcg MPER-656 mo(0,2,6,12) (N=15) | Control 1: Placebo for MPER-656 mo(0,2,6,12) (N=1) | Control 2: Placebo for MPER-656 mo(0,2,6,12) (N=3)
Any Event in SOC (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 1 (1) | 8 (8) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT03934541/Prot_SAP_002.pdf
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03934541/ICF_001.pdf